CLINICAL TRIAL: NCT04000698
Title: A Phase I-II Pilot Clinical Trial of Safety and Efficacy of Personalized Targeted Preparative Regimen With Allogeneic TcRαβ/CD19-depleted Hematopoietic Stem Cell Transplantation and Posttransplant Donor T- Cells Infusion in Children With Chemoresistаnt Acute Leukemia.
Brief Title: Personalized Targeted Preparative Regimen Before T-depleted Allogeneic HSCT in Children With Chemoresistent Acute Leukemias
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCPHOI-2018-08
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Refractory Acute Myeloid Leukemia; Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention/treatment (Experimental): Preparative chemotherapy before allogeneic HSCT
  * Fludarabin
  * Cytarabine
  * Venetoclax
  * Daratumomab
  * Vecanoid
  * treosulfan
  * fludarabine
  * thiophosphomide
  * Venetoclax
  * Plerixafor
  * abatacept
  * tocilizumab
  * rituximab
  * HSCT from the haploidentical donor, ex vivo depleted of alpha/beta T lymphocytes
  Interventions: Drug: Preparative regimen

INTERVENTIONS:
Drug: Preparative regimen — Preparative chemotherapy before allogeneic HSCT
  * Fludarabin
  * Cytarabine
  * Venetoclax
  * Daratumomab
  * Vecanoid Condition
  * treosulfan
  * fludarabine
  * thiophosphomide
  * Venetoclax
  * Plerixafor GVHD prophylaxis
  * abatacept
  * tocilizumab
  * rituximab
  * HSCT from the haploidentical donor, ex vivo depleted of alpha/beta T lymphocytes

SUMMARY:
The purpose of this study is to evaluate the safety and efficiency of personalized targeted therapy in combination with high-dose chemotherapy as part of a preparative regimen before T-depleted allogeneic hematopoietic stem cell transplantation in children with chemoresistant acute leukemias

DETAILED DESCRIPTION:
The outcome of hematopoietic stem cell transplantation (HSCT) in a cohort of children with chemorefractory leukemia is poor. The incidence of relapse exceeds 50% and survival varies from 10 to 40%. Additional attempts at remission induction with various combinations of chemotherapy are unlikely to improve the outcome and will contribute to toxicity.

The hypothesis of the study is that personalized targeted therapy combined with high-dose chemotherapy may improve the outcome of allogeneic HSCT in a cohort of pediatric patients with refractory leukemia.

Bcl-2, CD38, CD184 were chosen as potential targets due to frequent expression in pediatric acute leukemias, availability of marketed targeted therapies venetoclax, daratumumab and prelixafor, and expected non-overlapping toxicity profile of these agents and the conditioning regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent (for patients > 14 years old). For subjects < 18 years old their legal guardian must give informed consent
2. Disease stage

   * Acute myeloid leukemia (AML), relapsed or refractory, failure to achieve hematologic remission after at least to courses of intensive chemotherapy, including at least one course with high-dose AraC and fludarabine
   * Acute lymphoblastic leukemia (ALL), relapsed or refractory, failure to achieve hematologic remission after at least two high-dose therapy blocks
3. Patient eligible for current hematopoietic stem cell transplantation protocol
4. The BCL-2 expression must be detected on greater than 30% of tumor cells (AML and ALL) by flow cytometry
5. CD38 expression must be detected on greater than 30% of tumor cells (AML and ALL) by flow cytometry
6. CD184
7. Patients must have measurable or evaluable disease at the time of enrollment, which may include any evidence of disease including minimal residual disease detected by flow cytometry, cytogenetics, or polymerase chain reaction (PCR) analysis.
8. Patient Clinical Performance Status: Karnofsky >50% or Lansky >50%
9. Patient Life Expectancy >12 weeks
10. Patients who agree to long-term follow up for up to 5 years

Exclusion Criteria:

* Age >25 years
* Patients with uncontrolled infections
* Clearance of creatinine < 70 ml/min
* Cardiac ejection fraction < 40%
* Patients who can perform pulmonary function tests will be excluded if they have a diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin) of < 50% predicted; patients who are unable to perform pulmonary function tests will be excluded if the oxygen (O2) saturation is < 92% on room air
* Patients who have liver function test (LFTs) (including total bilirubin, aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) >= twice the upper limit of normal
* Karnofsky/Lansky Scale <70%

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence of neutrophil and platelets engraftment at day +30 after HSCT | 30 days after HSCT
Overall response rate | 30 days after HSCT
  Proportion of patients with hematologic remission at time points
Partial response rate | 30 days after HSCT
  Proportion of patients with MRD negativity at time points
Rate of toxicity stage > 3 according to CTCAE 5.0 | 40 days after first drug administration
  Proportion of patients with allergic/ anaphylaxis reaction toxicity stage > 3 according to CTCAE 5.0
cumulative incidence of transplant-related mortality | 100 days after HSCT

SECONDARY OUTCOMES:
Rate of expression of target molecule on blast cells | 1 week before first drug administration
  Proportion of patients with target molecule on blast cells: CD38 and/or CD 184 and/or Bcl2
cumulative incidence of acute GVHD grade II-IV | 120 days after HSCT
cumulative incidence of chronic GvHD | 1 year after HSCT
Rate of immune recovery at day 30 | 30
  Proportion of patients with early immune recovery: T-cell, NK- cell, B-cell >determined numbers
overall survival | 1 year after HSCT
event-free survival | 1 year after HSCT

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia